CLINICAL TRIAL: NCT02696863
Title: Plan for Systematic Identification of Lung Cancers of Occupational Origin: Implementation Study
Acronym: RECAP 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-05
Record Dates: First submitted 2016-02-08; First posted 2016-03-02 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Broncho Pulmonary Cancer
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- filling a questionnaire and interview: The questionnaire is tracking occupational carcinogens. It consists of 30 questions , fills an average of 3 minutes and includes three response categories: "yes", "no" and "do not know". A questionnaire will be added social and professional issues.
  Interviews will be conducted with the patient to identify obstacles and facilitating elements
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire

SUMMARY:
The main objective is to identify obstacles and elements facilitating the implementation of a tracking device Broncho Pulmonary Cancer during the course of care.

The secondary objective is to assess patient knowledge and information received on their previous occupational exposure during their professional activity.

This is a prospective multicenter study of qualitative methodology through in-depth interviews conducted with patients treated at ICLN and CHU Saint-Etienne

ELIGIBILITY:
Inclusion Criteria:

* primitive CBP Patients;
* Patients employees or have been employees of the general scheme and / or the agricultural social security system;
* Patients understand French.

Exclusion Criteria:

* Patients recognized occupational disease for CBP;
* recognized disability in patients for CBP by the social security system;
* Patients who have never been employees of the General or the agricultural social security system plan
* Patients already included in phase 1 of the study;
* Refusal of participation, signed consent major patients protected under guardianship;
* Patients unable to understand the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primitive CBP Patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Interview | 45 minutes
  Obstacles and elements facilitating the establishment of a work-related bronchopulmonary cancer tracking device during the course of care. These are collected in an interview with a sociologist. It will be analyse with NVivo.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Saint-Etienne, Saint-Etienne
  - ICLN, Saint-Priest-en-Jarez